CLINICAL TRIAL: NCT07398001
Title: Discontinuation of Antiplatelet Therapy After Drug-Coated Balloon Treatment
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ulsan University Hospital (Other)
Responsible Party: Principal Investigator, Eun-Seok Shin, Professor, Ulsan University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025-04-042
Record Dates: First submitted 2026-01-20; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Percutaneous Coronary Intervention; Antiplatelet Therapy; Drug-coated Balloon
Keywords: coronary artery disease; drug-coated balloon; percutaneous coronary intervention; antiplatelet therapy; clinical outcomes
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stop Antiplatelet (Experimental): Antiplatelet discontinuation group
  Interventions: Drug: Stop Antiplatelet
- Continue Antiplatelet (Active Comparator): Antiplatelet continuation group
  Interventions: Drug: Continue Antiplatelet

INTERVENTIONS:
Drug: Stop Antiplatelet — Antiplatelet discontinuation after DCB treatment
  Arms: Stop Antiplatelet
Drug: Continue Antiplatelet — Antiplatelet continuation after DCB treatment
  Arms: Continue Antiplatelet

SUMMARY:
The goal of this clinical trial is to evaluate the benefits and risks of discontinuing antiplatelet therapy on clinical outcomes in patients who previously underwent coronary intervention using a drug-coated balloon.

The main questions it aims to answer are:

Does stopping antiplatelet therapy after 12 months affect the risk of net adverse clinical events? Does stopping antiplatelet therapy reduce the risk of bleeding compared with continuing treatment?

Researchers will compare patients who discontinue antiplatelet therapy with patients who continue antiplatelet therapy to determine the impact on clinical outcomes during follow-up.

Participants will:

Be randomly assigned to either discontinue or continue antiplatelet therapy Receive routine clinical follow-up through clinic visits or telephone contacts Be monitored for cardiovascular events and bleeding outcomes over time

DETAILED DESCRIPTION:
Coronary artery disease is a major cause of morbidity and mortality worldwide. Percutaneous coronary intervention is widely used for the treatment of coronary artery disease, traditionally involving implantation of drug-eluting stents. Although contemporary drug-eluting stents have improved safety and efficacy compared with earlier stent technologies, permanent metallic implants remain associated with long-term considerations, including restenosis, stent thrombosis, and the need for prolonged antiplatelet therapy.

Drug-coated balloon therapy represents an alternative revascularization strategy that delivers an antiproliferative drug to the coronary vessel wall without implantation of a permanent scaffold. This "leave-nothing-behind" approach has been adopted in specific clinical settings and has been increasingly applied in selected coronary lesions. The absence of a permanent implant may offer potential advantages with respect to long-term vessel healing and antiplatelet therapy management.

Bleeding complications after coronary intervention are clinically relevant and have been associated with adverse outcomes. Decisions regarding the duration of antiplatelet therapy require careful consideration of both ischemic and bleeding risks. While shorter durations of antiplatelet therapy have been explored following contemporary coronary interventions, optimal long-term antiplatelet strategies after drug-coated balloon-based procedures remain incompletely defined.

Limited data are available regarding the clinical outcomes associated with discontinuation of antiplatelet therapy beyond 12 months in patients who have undergone initial percutaneous coronary intervention using drug-coated balloon treatment and have remained clinically stable. As a result, uncertainty persists regarding the balance of potential benefits and risks of long-term antiplatelet therapy in this population.

This prospective, randomized, multicenter study is designed to compare clinical outcomes between patients who discontinue antiplatelet therapy and those who continue antiplatelet therapy after 12 months following drug-coated balloon-based percutaneous coronary intervention. The study aims to provide additional evidence to inform clinical decision-making regarding antiplatelet therapy management in patients treated with drug-coated balloons.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged 19 years or older who are able to understand the risks, benefits, and treatment alternatives of the study and who provide written informed consent voluntarily.
2. Patients who underwent drug-coated balloon treatment at least 12 months prior to enrollment.
3. Patients who have not experienced major adverse cardiovascular events, including myocardial infarction, stroke, or target vessel revascularization, since the index DCB treatment.
4. Patients who have not experienced major bleeding since the index DCB treatment.
5. Patients who are receiving antiplatelet therapy at the time of enrollment.

Exclusion Criteria:

1. Patients with concomitant vascular disease requiring long-term antiplatelet therapy.
2. Patients with non-cardiac comorbid conditions that, in the judgment of the investigator, are associated with a life expectancy of less than 1 year or may result in poor compliance with the study protocol.
3. Patients who are participating in another drug or coronary device clinical study at the time of enrollment.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1042 (Estimated)
Dates: Start 2026-02-12 (Estimated); Primary Completion 2028-02-11 (Estimated); Study Completion 2030-07-31 (Estimated)

PRIMARY OUTCOMES:
Net adverse clinical events (NACE) | Up to 12 months after randomization
  A composite of all-cause death, non-fatal myocardial infarction, clinically driven target vessel revascularization, and bleeding defined as Bleeding Academic Research Consortium (BARC) type 2 to 5.
  Non-fatal myocardial infarction is defined as a myocardial infarction diagnosed using standard clinical, electrocardiographic, and biomarker criteria that does not result in death.

SECONDARY OUTCOMES:
NACE | Up to 24, 36 months after randomization
  A composite of all-cause death, non-fatal myocardial infarction, clinically driven target vessel revascularization, and bleeding defined as Bleeding Academic Research Consortium (BARC) type 2 to 5.
The single components of the primary endpoint | Up to 12, 24, 36 months after randomization
  A composite of all-cause death, non-fatal myocardial infarction, clinically driven target vessel revascularization, and bleeding defined as Bleeding Academic Research Consortium (BARC) type 2 to 5.
Rate of cardiac death | Up to 12, 24, 36 months after randomization
  Cardiac death is defined as death resulting from an immediate cardiac cause, including myocardial infarction, heart failure, fatal arrhythmia, or sudden cardiac death. Deaths of unknown cause or unwitnessed deaths without an identifiable non-cardiac cause are also classified as cardiac death. Deaths clearly attributable to non-cardiac causes, such as malignancy, infection, trauma, or other non-cardiovascular conditions, are not considered cardiac death.
Stroke (ischemic and hemorrhagic) | Up to 12, 24, 36 months after randomization
  Stroke is defined as a new, sudden onset of a focal or global neurological deficit lasting 24 hours or longer, or resulting in death, with a vascular cause. Both ischemic stroke and hemorrhagic stroke are included. The diagnosis is confirmed by clinical assessment and supported by brain imaging when available. Transient ischemic attacks (TIA), defined as neurological symptoms resolving within 24 hours without evidence of infarction or hemorrhage, are not considered stroke.
Target lesion failure | Up to 12, 24, 36 months after randomization
  A composite of cardiac death, target vessel-related myocardial infarction, or clinically indicated target lesion revascularization.
Angina severity measured with Seattle Angina Questionnaires | At baseline and 12 months after randomization
  Angina severity is assessed using the Seattle Angina Questionnaire (SAQ), a validated, patient-reported questionnaire designed to measure the impact of angina on daily life. The questionnaire evaluates angina-related symptoms, physical limitation, and quality of life. Higher scores indicate fewer angina symptoms and better functional status. Changes in SAQ scores over time are used to assess angina severity during follow-up.
Cost-effectiveness | Up to 12, 24, 36 months after randomization
  Cost-effectiveness is defined as an economic evaluation comparing the costs and clinical outcomes of the study treatment strategies. Direct medical costs related to treatment, follow-up care, hospitalizations, and management of clinical events are assessed and compared in relation to clinical outcomes during the follow-up period. Cost-effectiveness is evaluated to determine the relative economic value of discontinuing versus continuing antiplatelet therapy.
Sex difference in NACE | Up to 12, 24, 36 months after randomization
  Sex differences are assessed by comparing the incidence of NACE between male and female participants during follow-up.
Comparison of NACE in DM patients | Up to 12, 24, 36 months after randomization
  NACE in patients with diabetes mellitus is assessed as a composite of ischemic and bleeding events during follow-up after randomization.
NACE in patients with acute coronary syndrome | Up to 12, 24, 36 months after randomization
  Acute coronary syndrome was defined as ST-segment elevation myocardial infarction, non-ST-segment elevation myocardial infarction, or unstable angina.

CONTACTS AND LOCATIONS:
Locations (7):
- South Korea (7):
  - Korea University Ansan Hospital, Ansan
  - Kangwon National University Hospital, Chuncheon
  - Kosin University Hospital, Pusan
  - Korea University Guro Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Ulsan Medical Center, Ulsan
  - Ulsan University Hospital, Ulsan

IPD SHARING:
Plan to Share IPD: Yes
Only de-identified individual participant data necessary to reproduce the main analyses will be shared. Data sharing will be subject to approval of a research proposal and execution of a data use agreement.
Time Frame: Beginning 6 months after publication of the primary results and ending 5 years thereafter.
Access Criteria: Researchers who provide a methodologically sound research proposal may request access to the de-identified individual participant data. Requests will be reviewed by the study steering committee, and access will be granted following approval of the proposal and execution of a data use agreement.